CLINICAL TRIAL: NCT06518278
Title: Assessing Central Nervous System Contributions to Accelerate Musculoskeletal Pain Diagnosis and Treatment
Brief Title: Assessing Central Aspects of Pain
Acronym: AsCent
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other); Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 24030; Versus Arthritis (Other Grant/Funding Number: 23145); EULAR (Other Grant/Funding Number: 1016807)
Record Dates: First submitted 2024-06-13; First posted 2024-07-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis; Fibromyalgia; Chronic Low Back Pain; Inflammatory Arthritis
Keywords: Quantitative Sensory Testing; Temporal Summation; Pressure Pain detection Threshold; Conditioned Pain Modulation; Offset Analgesia
MeSH Terms: conditions — Osteoarthritis; Fibromyalgia; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal Pain: Adults aged 18 years or older self-reporting one or more of the following: Osteoarthritis, Fibromyalgia, Chronic Low Back Pain, Inflammatory Arthritis and pain of >3/10 for most days in the past 3 months before baseline.

SUMMARY:
BACKGROUND: Chronic pain continues for more than 12 weeks despite medication or treatment. Chronic pain is the main symptom of muscle and joint problems, rarely explained by damage to the muscle and joints alone. Activity in the central nervous system (CNS; nerves, spinal cord, and brain) pathways governs our ability to describe pain intensity and our emotional response to pain. Musculoskeletal conditions (e.g., inflammatory arthritis, osteoarthritis, low back pain, fibromyalgia) share altered CNS pathways, acknowledged by recent classifications of 'primary' and 'nociplastic' pain. Clinically useful tools to diagnose and measure activity and reveal abnormalities in these CNS pathways are needed to improve clinical decisions and accelerate new treatment development. Laboratory pain sensitivity testing and brain imaging confirm the CNS as a primary contributor to pain. These assessments are less acceptable or unfeasible for clinical practice. Simpler clinical pain sensitivity assessments are being developed. The investigators simple Central Aspects of Pain (CAP) questionnaire detects some people with pain sensitivity and knee, rheumatoid arthritis or low back pain. Combining the CAP questionnaire reflecting emotional processing and simpler pain sensitivity assessment, combining two different dimensions should be better than either approach alone.

PURPOSE: To optimise diagnosis and measurement of CNS as the primary contribution to chronic musculoskeletal pain by using the CAP questionnaire and simpler pain sensitivity assessments to ensure timely, effective diagnosis and treatment.

OBJECTIVES: 1. Assess the ease, ability and performance of the combined CAP questionnaire and simpler pain sensitivity assessments to identify CNS as the primary contributor to chronic pain across musculoskeletal conditions.

2. Use the CAP questionnaire alone or with substitute measures of activity in CNS pathways, demographic, and clinical variables to indicate pain levels at six and twelve weeks.

3. Understand the relationship between CAP and simpler pain sensitivity assessment with laboratory pain sensitivity assessments as a tool to inform the current CNS activity contributing to pain.

4. Evaluate associations between the CAP questionnaire and simpler pain sensitivity assessments with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or over.
* One for more of the following self-reported diagnoses: fibromyalgia, inflammatory MSK condition (e.g., rheumatoid arthritis, psoriatic arthritis, axial spondyloarthritis), low back pain, osteoarthritis.
* MSK diagnosis and pain onset more than 3 months prior to baseline
* Self-reported pain levels ≥ 3 on a 0 to 10 numerical rating scale where 0 = 'no pain' and 10 = 'worst pain imaginable' on most days in the 3 months before baseline.
* Ability to give informed consent.

Exclusion Criteria:

* Terminal/uncontrolled medical or mental health condition that would prevent participants from completing assessments or pose a significant risk to participants or staff.
* Insufficient understanding of spoken or written English to comply with the requirements of the study protocol.
* Inability to adhere to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include people with musculoskeletal pain attending NHS outpatient clinics and individuals who have consented to be contacted for future research from research databases at the University of Nottingham
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Central Aspects of Pain Questionnaire | Baseline, 6 and 12 weeks
  Zero indicates low levels of central aspects of pain, 16 indicated high central aspects of pain
Simpler pain sensitivity measures | Baseline
  Simpler pain sensitivity will be assessed as a combination of the point at pressure changes from a feeling of pressure to a feeling of pain or discomfort (kg), temporal summation is measured at the difference between one stimuli and ten consecutive stimuli scores from 0-10 of a Visual Analog Scale (0 = no pain or sharpness, 10 = worse pain or sharpness). Conditioned pain modulation will assess the point at which pressure changes to pain or discomfort (kg) when a conditioned stimuli is applied to the contralateral arm. The number of tender sites will be assessed by palpating 18 body sites and scored based on the number of tender sites reported. Conditioned pain modulation will also be assessed based on the number of tender sites reported with and without a conditioned stimuli to the forearm. Low scores indicate low pain sensitivity, high scores indicate high pain sensitivity.

SECONDARY OUTCOMES:
Sleep efficiency | Baseline
  Time difference between total sleep time and time in bed (total sleep time/time in bed) zero is poor sleep efficiency, 1 is the best sleep efficiency
Hospital Anxiety and Depression Scale (HADs) | Baseline, 6 and 12 weeks
  0 is normal levels of anxiety or depression, 21 abnormal (case) of anxiety or depression
Central Sensitization Index (CSI) | Baseline, 6 and 12 weeks
  scored from 0-36 higher scores indicating greater central sensitisation severity
McGill pain | Baseline, 6 and 12 weeks
  0 (no pain) to 78 (severe pain)
Self-reported Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (S-LANSS) | Baseline, 6 and 12 weeks
  Scored 0-21. Scoring a score of 12 or more suggests pain of predominantly neuropathic origin
Fibromyalgia classification criteria | Baseline, 6 and 12 weeks
  Fibromyalgia classification criteria presence of fibromyalgia determined based on a combined score from the widespread pain index (WPI) ≥7 and symptom severity (SS) scale score ≥5 or WPI 3 - 6 and SS scale score ≥9
Cognitive Failures Questionnaire (CFQ) | Baseline, 6 and 12 weeks
  Scores range from 0-100. A higher total score indicates more subjective cognitive failure.
Health Assessment Questionnaire (HAQ) | Baseline, 6 and 12 weeks
  The score goes from 0 (no incapacity) to 3 (full incapacity); a score below 0.5 is considered normal whereas a score above 1.5 indicates severe disability.
Fatigue Impact Scale (FIS) | Baseline, 6 and 12 weeks
  Scores range from 0 (No problem) to 160 (extreme problems)
36-Item Short Form Survey (SF-36) | Baseline, 6 and 12 weeks
  Score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Pittsburgh Sleep Quality (PSQI) | Baseline, 6 and 12 weeks
  Global PSQI score, which ranges from 0 to 21. A global PSQI score over 5 indicates poor sleep relative to clinical and laboratory measures, and higher scores indicate poorer sleep quality
Laboratory pain sensitivity | Baseline
  Laboratory pain sensitivity will be assessed as a combination of the point at pressure changes from a feeling of pressure to a feeling of pain or discomfort (kPa), temporal summation is measured at the difference between one stimuli and ten consecutive stimuli scores from 0-10 of a Visual Analog Scale (0 = no pain or sharpness, 10 = worse pain or sharpness). Conditioned pain modulation will assess the point at which pressure changes to pain or discomfort (kPa) when a conditioned stimuli is applied to the contralateral arm. Heat pain threshold is the temperature (degrees) at which the feeling of heat changes to one of pain or discomfort. Offset analgesia is the difference in visual analog pain scores (0 = no pain) 10 = worst imaginable pain) from the temperature at time point 1 and the temperature at time point 3.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Academic Rheumatology, IRIS, School of Medicine, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pre-planned analyses will be performed by the study team. Requests for collaborative analyses of IPD, using non-identifiable data, may be made to the study PI and through Alleviate data hub.